CLINICAL TRIAL: NCT05383950
Title: Rehabilitation of Chronic Diseases and Smart Health Management System Service Provided by Hospital and Community Association
Brief Title: Rehabilitation of Chronic Diseases and Smart Health Management System Service
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0562
Record Dates: First submitted 2022-05-01; First posted 2022-05-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Rehabilitation; Cardiac Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- smartphone application based 12-week pulmonary or cardiac rehabilitation (Experimental)
  Interventions: Device: smartphone application

INTERVENTIONS:
Device: smartphone application — In this study, the investigators will provide smartphone application based 12-week pulmonary or cardiac rehabilitation program to patients with chronic respiratory, cardiac, or geriatric diseases.

SUMMARY:
In Republic of Korea, it is not easy to practice standard pulmonary rehabilitation (PR) or cardiac rehabilitation (CR). In this study, the investigators will provide newly developed smartphone application to patients with chronic respiratory, cardiac, or geriatric diseases. The investigators want to confirm whether participants, who perform smartphone application based 12-week PR or CR program, present improved exercise capacity, dyspnea symptom, muscle strength, or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea symptom >= mMRC 1 or NYHA I
* adults between 20 years and 80 or years

Chronic respiratory disease

* FEV1/FVC < 0.7 in pulmonary function test
* bronchiectasis in more than one lobe on chest computed tomography
* FVC of DLCO < 0.8 of predicted value in pulmonary function test

Chronic cardiac disease

* Reperfusion Therapy for angina pectoris or myocardial infarction
* Heart failure with reduced ejection fraction (LVEF < 50%)

Chronic geriatric disease

* Ages between 60 and 80 years
* Clinical frailty scale between 1 and 4

Exclusion Criteria:

* history of acute exacerbation within 4 weeks
* unable to comply rehabilitation program
* not suitable for study on decision by duty physician
* no consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change of 6 minutes walk distance at 12 weeks (Chronic respiratory disease group) | 12 weeks
  The distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
change of maximal oxygen consumption (VO2max) at 12 weeks (Chronic respiratory disease group, Chronic cardiac disease group) | 12 weeks
  The maximum rate of oxygen consumption measured during incremental exercise test (cardiopulmonary exercise test).
change of frailty index at 12 weeks (Chronic geriatric disease group) | 12 weeks
  The frailty index is defined as the proportion of deficits present in an individual out of the total number of age-related health variables considered.
  Frailty Index (FI) = (number of health deficits present) ÷ (number of health deficits measured)
  For example, a person with 20 of 40 deficits collected has an FI score of 20/40 = 0.5
  The frailty index ranges 0 (best performance) to 1 (worst performance).

SECONDARY OUTCOMES:
change from dyspnea symptom at 12 weeks (Chronic respiratory disease group, Chronic geriatric disease group) | 12 weeks
  Dyspnea symptom is measured according to the Modified Medical Research Council (mMRC) Dyspnea Scale.
  The mMRC scale is from 0 to 4:
  0, no breathlessness except on strenuous exercise
  1. shortness of breath when hurrying on the level or walking up a slight hill
  2. walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level
  3. stops for breath after walking ∼100 m or after few minutes on the level
  4. too breathless to leave the house, or breathless when dressing or undressing
change from dyspnea symptom at 12 weeks (Chronic cardiac disease group, Chronic geriatric disease group) | 12 weeks
  Dyspnea symptom is measured according to the New York Heart Association Functional Classification (NYHA class).
  The NYHA class is from I to IV:
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation (feeling heart beats), or dyspnea (shortness of breath).
  Class II(Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III(Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV(Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
Change of EuroQol 5-dimension 5-level (EQ-5D-5L) score at 12 weeks (all groups) | 12 weeks
  A questionnaire assessing health related quality of life on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each item is scored 1-5, yielding a total between 5 and 25.
  The scores range from 5 (best performance) to 25 (worst performance).
change of Korean Health-related Quality of Life Instrument with 8 Items (HINT-8) score at 12 weeks (all groups) | 12 weeks
  A questionnaire assessing health related quality of life on 4 health dimensions (physical, mental, social, positive health dimension). Each item is scored 1-4, yielding a total between 8 and 40.
  The scores range from 8 (best performance) to 40 (worst performance).
change of muscle strength at 12 weeks (all groups) | 12 weeks
  The muscle strength measures hand grip strength. The cut-off value for sarcopenia is < 30 kg
change of Short physical performance battery (SPPB) at 12 weeks (all groups) | 12 weeks
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons.
  The scores range from 0 (worst performance) to 12 (best performance). The cut off value for sarcopenia is ≤ 8.
change of muscle mass at 12 weeks (all groups) | 12 weeks
  The muscle mass is measured using the Bioelectrical Impedance Analysis. The cut off value for sarcopenia is < 7.26 kg/m^2.
change of forced expiratory volume in one second (FEV1) at 12 weeks (Chronic respiratory disease group) | 12 weeks
  The forced expiratory volume in one second (FEV1) is measured using spirometry. The value will be presented in % predicted value.
change of forced vital capacity (FVC) at 12 weeks (Chronic respiratory disease group) | 12 weeks
  The forced vital capacity (FVC) is measured using spirometry. The value will be presented in % predicted value.
change of diffusing capacity of the lung for carbon monoxide (DLCO) at 12 weeks (Chronic respiratory disease group) | 12 weeks
  The diffusing capacity of the lung for carbon monoxide (DLCO) is measured using single breath holding method.
  The value will be presented in % predicted value.
Change of chest pain symptom at 12 weeks (Chronic cardiac disease group) | 12 weeks
  Chest pain symptom is measured according to the Canadian Cardiovascular Society grading of angina pectoris (CCS angina grade).
  The CCS angina grade is from I to IV:
  Grade I: Angina with strenuous/rapid/prolonged exertion at work or recreation only; no angina with ordinary physical activity, e.g. walking, climbing stairs Grade II: Ordinary activity slightly limited: angina with walking/climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold/wind, under emotional stress, during few hours after awakening, walking >2 blocks on level ground, or climbing >1 flight of stairs at normal pace and normal conditions Grade III: Marked limitation of ordinary physical activity: angina with walking 1-2 blocks on level ground or climbing 1 flight of stairs at normal pace and normal conditions Grade IV: Inability to carry on any physical activity without discomfort; anginal syndrome may be present at rest
change of exercise duration in cardiopulmonary exercise test at 12 weeks (Chronic cardiac disease group) | 12 weeks
  This test measures total exercise duration.
change of exercise capacity in cardiopulmonary exercise test at 12 weeks (Chronic cardiac disease group) | 12 weeks
  This test measures metabolic equivalents (METs).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chung C, Kim AR, Kim D, Kwon H, Lee SH, Jang IY, Jo MW, Kang DY, Lee SW. Smartphone application-based rehabilitation in patients with chronic respiratory and cardiovascular diseases. Sci Rep. 2024 Feb 6;14(1):3018. doi: 10.1038/s41598-024-53583-2. PMID 38321153